CLINICAL TRIAL: NCT01640860
Title: A Phase II Study of Concurrent Chemoradiotherapy With Weekly Docetaxel and Cisplatin in Inoperable Esophageal Cancer
Brief Title: Concurrent Chemoradiotherapy With Docetaxel and Cisplatin in Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Sang-Hee Cho, professor, Chonnam National University Hospital
Other Study IDs: DCESO; CUNHH (Other: CNUHH)
Record Dates: First submitted 2008-01-07; First posted 2012-07-16 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Cancer
Keywords: docetaxel; cisplatin; combined modality therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to determined the feasibility and safety in advanced esophageal cancer treated with docetaxel and cisplatin cocurrent chemoradiotherapy. The primary end points were clinical best response and response rate and secondary endpoints were progression free survival and overall survival.

DETAILED DESCRIPTION:
Chemotherapy can provide significant palliation of symptoms for patients with unresectable, locally advanced or metastatic esophageal cancer. Cisplatin and continuous infusion 5 FU, alone or combined with radiotherapy, is the most frequently used regimen. The response rate reported with cisplatin and 5 FU ranged from 35 to 40% ,whereas the 2-year survival rates of patients with locally advanced esophageal cancer ranged from 8 to 55%, with a mean 27%. Therefore, there is a need to test new combination, specifically in unresectable locally advanced esophageal patients, with the aim of increasing the pCR rate and survival. Cisplatin had been widely used as radiosensitizer and Docetaxel is different from that of cisplatin -5FU and and has proved to have an additive effect with cisplatin and supra-additive antitumor activity with fluorouracil in vitro and in murine models. To investigate the feasibility of combining concomitant radiation with docetaxel and cisplatin and assess the regimen's toxicity, locoregional control rate, and survival in patients with locally advanced or metastatic esophageal cancer.In this study, docetaxel 25mg/m2 is given with 500ml normal saline , as a 1hr infusion, on days 1,8 of every 3 weeks. Cisplatin75mg/m2 is given by intravenous infusion in 500 mL of 5% dextrose solution over 60 minutes on day 1 of every 3weeks.. Therapy will be repeated every 21 days. Radiation therapy (200cGy/day upto 5400 cGy) begin on the first day of week 1 over 6 weeks (concomitant chemoradiation therapy). When the investigators assume that standard treatment's response rate is 50% and the response of experimental treatment is 75% and use Simon's two-stage optimal design under the significance level of 5% and the power of 80%, the total sample size of 25 is at least required. For a total of 25 subjects, 11 will be accrued during stage 1 and 14 during stage 2. If 6 or fewer responses are observed during the first stage then the trial is stopped early. If 16 or fewer responses are observed by the end of the trial then no further investigation of the drug is warranted. If the investigators assumed that the drop out rate was 10%, number of subjects per treatment arm will be 28.

ELIGIBILITY:
Inclusion Criteria:

1. 18<age<75 years
2. histologically proven and previously untreated SCC of the esophagus
3. WHO performance status(PS)≤2
4. absolute neutrophil count≥2,000/uL, platelet count≥100,000/uL
5. adequate renal and hepatic function
6. No prior chemotherapy but prior adjuvant chemotherapy finished at least 6 months before enrollment was allowed
7. No prior radiation therapy for at least 4 weeks before enrollment in the study

Exclusion Criteria:

1. Evidence of distant metastases
2. Pleural of pericardial effusion
3. Fistulisation
4. Prior malignancies(other than basal cell skin carcinoma)
5. Prior myocardial infarction or uncontrolled infection
6. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
7. History of significant neurologic or psychiatric disorders including dementia or seizures
8. Other serious underlying medical conditions which could impair the ability of the patient to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced esophageal cancer diagosed at Chonnam National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 4-6 weeks after completion of CRT
  Chest and abdominal CT and EGD were obtained to assess tumor status, 4 to 6 weeks after the completion of CRT. The patients who were documented on the CT scan and upper gastrofibroscopy as showing a complete response (CR) underwent positron emission tomography (PET)-CT. If the PET-CT showed no metabolic evidence of malignancy, we deemed the response to be a CR.

SECONDARY OUTCOMES:
progression free survival, overall survival and adverse events | every 3-6 months
  Tumor resection with extended en bloc lymphadenectomy was performed in operable patients approximately 4 to 8 weeks after treatment. Follow-up evaluation was performed every 3months for the first 2years, then every 6monhs for the next 3 years, then annually until patinet death or loss to follow-up. This included clinical examination, dysphagia score, assessment of late radiation toxicity and repeat CT scan of chest/ abdomen and EGD.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hee Cho, MD. PhD, Principal Investigator — CNUHH
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeolanamdo, South Korea